CLINICAL TRIAL: NCT06910059
Title: The CT-verified Data Collection Study to Investigate the Correlation Between the Leadless Pacemaker Tip Location and Echo, ECG
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Micra-CT EM Study
Record Dates: First submitted 2025-03-14; First posted 2025-04-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Bradycardia Sinus; AV Block; Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrioventricular Block; Atrial Fibrillation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational — It is a observational study and patients with pacing indications who plan to receive Micra AV implantation will be recruited. No intervention procedure will be performed.

SUMMARY:
The goal of this observational study is to assess inter-/intra- ventricular synchrony and ECG characteristics in relation to Micra tip location.

The secondary objective is (1) to identify an optimal Micra pacing location to improve LV function, (2) to investigate the correlation between Micra tip location and tricuspid regurgitation, and (3) to investigate whether Micra location would impact AV synchrony. Patients with pacing indications who plan to receive Micra AV implantation will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years old
* Patients who are willing to provide Informed Consent
* Patients with Class I or II indications who plan to receive a leadless pacemaker, including SSS, AVB, AF with bradycardia, etc.
* Patients who plan to conduct a cardiac CT scan after implantation

Exclusion Criteria:

* Patients with lead retention
* Patients had heart valve replacement
* Patients diagnosed with ischemic heart diseases
* Patients who are allergic to or refuse to use contrast in CT scans
* Patients who are pregnant or have a plan for pregnancy during the study
* Patients with medical conditions that would limit study participation
* Patients already enrolled in another clinical trial which would impact participation of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 40 subjects in site. Patients with pacing indications who plan to receive Micra AV implantation will be selected.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of ECG characteristics in relation to Micra tip location | Within 6 months after the surgery.
  Patients' ECG will be measured to see whether there is difference in ECG characteristics between Micra tip locations.

SECONDARY OUTCOMES:
Cardiac functional changes | Within 6 months after the surgery.
  LVEF, RV length and quantity of tricuspid regurgitation will be measured.
To investigate whether Micra location would impact AV synchrony | Within 6 months after the surgery.
  Percentage of AV synchrony will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds D, Duray GZ, Omar R, Soejima K, Neuzil P, Zhang S, Narasimhan C, Steinwender C, Brugada J, Lloyd M, Roberts PR, Sagi V, Hummel J, Bongiorni MG, Knops RE, Ellis CR, Gornick CC, Bernabei MA, Laager V, Stromberg K, Williams ER, Hudnall JH, Ritter P; Micra Transcatheter Pacing Study Group. A Leadless Intracardiac Transcatheter Pacing System. N Engl J Med. 2016 Feb 11;374(6):533-41. doi: 10.1056/NEJMoa1511643. Epub 2015 Nov 9. PMID 26551877
- [Background] Udo EO, Zuithoff NP, van Hemel NM, de Cock CC, Hendriks T, Doevendans PA, Moons KG. Incidence and predictors of short- and long-term complications in pacemaker therapy: the FOLLOWPACE study. Heart Rhythm. 2012 May;9(5):728-35. doi: 10.1016/j.hrthm.2011.12.014. Epub 2011 Dec 17. PMID 22182495
- [Background] Kirkfeldt RE, Johansen JB, Nohr EA, Jorgensen OD, Nielsen JC. Complications after cardiac implantable electronic device implantations: an analysis of a complete, nationwide cohort in Denmark. Eur Heart J. 2014 May;35(18):1186-94. doi: 10.1093/eurheartj/eht511. Epub 2013 Dec 17. PMID 24347317